CLINICAL TRIAL: NCT01656434
Title: A Phase III, Randomized, Open-label, Active-controlled, Multicenter Trial to Study the Contraceptive Efficacy and Safety of the Commercial Batch of Oral Tablets of MK-8175A (Nomegestrol Acetate - 17ß-estradiol) in Healthy, Sexually-active Women Aged 18-50 Years
Brief Title: Study of the Contraceptive Efficacy and Safety of a NOMAC-E2 Combined Oral Contraceptive (COC)(P06448)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P06448; MK-8175A-022 (Other: Merck Protocol Number); SCH 900121 P06448 (Other: Merck Protocol ID)
Record Dates: First submitted 2012-07-31; First posted 2012-08-03 (Estimated); Results first posted 2015-03-17 (Estimated); Last update posted 2024-06-20 (Actual); Status verified 2022-02

CONDITIONS: Contraception
Keywords: Combined Oral Contraceptives
MeSH Terms: interventions — Ethinyl Estradiol; ferrous fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NOMAC-E2 (Experimental): Participants received a NOMAC-E2 tablet (2.5 mg nomegestrol acetate and 1.5 mg 17ß-estradiol), taken orally once daily for 13 cycles. Each cycle was 28 days. For each cycle, participants received NOMAC-E2 tablets on Days 1 to 24 and placebo tablets on Days 25 to 28.
  Interventions: Drug: NOMAC-E2; Other: Placebo
- NETA-EE (Active Comparator): Participants received a NETA-EE tablet (1 mg norethisterone acetate and 10 μg ethinylestradiol), taken orally once daily for 13 cycles. Each cycle was 28 days. For each cycle, participants received NETA-EE tablets on Days 1 to 24; EE 10 μg tablets on Days 25 and 26; and ferrous fumarate 75 mg tablets on Days 27 and 28.
  Interventions: Drug: NETA-EE; Drug: ethinylestradiol (EE); Drug: ferrous fumarate

INTERVENTIONS:
Drug: NOMAC-E2 — NOMAC-E2 film-coated oral tablets containing 2.5 mg nomegestrol acetate and 1.5 mg 17ß-estradiol.
  Other Names: MK-8175A; SCH 900121; Org 10486-0 (NOMAC); Org 2317 (E2)
  Arms: NOMAC-E2
Drug: NETA-EE — NETA-EE film-coated oral tablets containing 1 mg norethisterone acetate and 10 μg ethinylestradiol.
  Other Names: Lo Loestrin® Fe
  Arms: NETA-EE
Other: Placebo — tablet
  Arms: NOMAC-E2
Drug: ethinylestradiol (EE) — EE 10 μg tablet
  Arms: NETA-EE
Drug: ferrous fumarate — ferrous fumarate 75 mg tablet
  Arms: NETA-EE

SUMMARY:
The purpose of this study was to assess the contraceptive efficacy of a nomegestrol acetate + 17ß-estradiol (NOMAC-E2) combined oral contraceptive (COC) in healthy, sexually-active American women at risk for pregnancy. Vaginal bleeding patterns of women taking NOMAC-E2 were assessed and compared to those of women taking a norethisterone acetate + ethinyl estradiol (NETA-EE) COC. The safety of NOMAC-E2 was also assessed.

Participants were randomized to receive either NOMAC-E2 or NETA-EE in a 3:1 ratio. As of Amendment 1 (which increased the sample size of the NOMAC-E2 group), the randomization ratio was adapted accordingly for participants randomized after the sample size increase.

DETAILED DESCRIPTION:
This study was terminated early. The decision to terminate the study was based upon difficulties encountered with data collection (related to incomplete e-Diary entries) in concert with business considerations. The decision was not related to any new or unexpected safety or efficacy findings with NOMAC-E2. As a result of this early termination, none of the pre-specified efficacy endpoints were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Sexually active woman, at risk for pregnancy and in need of contraception
* Not planning to use other contraceptive methods (including barrier methods [e.g., condoms]) than the study drug, during the study
* Willing to use a COC for 12 months (13 cycles)
* Body mass index (BMI) of ≥18 and <38 kg/m^2
* Good physical and mental health
* Willing to complete an electronic diary on a daily basis for the duration of the study

Exclusion Criteria:

* Current smoker and age of >35 years
* Presence or history of either venous thromboembolic diseases (deep vein thrombosis [DVT], pulmonary embolism) or arterial thromboembolic diseases (myocardial infarction, stroke)
* History of migraine with focal neurological symptoms
* Diabetes mellitus with vascular involvement
* Less than two weeks of full remobilization from prolonged immobilization, major surgery, any surgery to the legs, or major trauma
* Severe hypertension
* Severe abnormal lipoproteins in the blood
* Pancreatic dysfunction
* Presence of history of severe liver disease or liver tumors
* Known or suspected sex steroid-influenced malignancies (e.g., of the genital organs or the breasts)
* Undiagnosed vaginal bleeding
* Known or suspected pregnancy
* Current or history of abuse of alcohol or drugs (e.g., laxatives)
* Abnormal cervical smear at screening
* Prior to start of treatment, spontaneous menstruation has not occurred following a delivery or abortion
* Breastfeeding or has been breastfeeding within 2 months prior to start of treatment
* Use of any investigational drugs and/or participation in any other clinical trial within 2 months prior to start of treatment
* Use of any of the following medications prior to or during the study may prohibit inclusion: sex hormones (other than pre- and post-treatment non-injectable contraceptives), injectable hormonal contraception, phenytoin, barbiturates, primidone, bosentan, carbamazepine, topiramate, felbamate, rifampicin, ritonavir, nevirapine, efavirenz, griseofulvin, herbal remedies containing Hypericum perforatum (e.g., St. John's wort)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3173 (Actual)
Dates: Start 2012-11-02 (Actual); Primary Completion 2014-02-12 (Actual); Study Completion 2014-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rolla E. Endometriosis: advances and controversies in classification, pathogenesis, diagnosis, and treatment. F1000Res. 2019 Apr 23;8:F1000 Faculty Rev-529. doi: 10.12688/f1000research.14817.1. eCollection 2019. PMID 31069056

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NOMAC-E2 | NETA-EE
Started | 2553 | 620
Treated | 2466 (One treated participant had incomplete data and was not included in the Safety Analyses.) | 604
Completed | 152 | 40
Not Completed | 2401 | 580
Not completed — Adverse Event | 199 | 63
Not completed — Enrollment terminated at trial site | 2 | 0
Not completed — Lost to Follow-up | 309 | 76
Not completed — Site discontinued study participation | 24 | 9
Not completed — Screen failure | 2 | 0
Not completed — Protocol Violation | 7 | 0
Not completed — Pregnancy wish | 18 | 6
Not completed — Pregnancy | 45 | 10
Not completed — Physician Decision | 7 | 2
Not completed — Non-compliance with study drug | 48 | 9
Not completed — Study terminated by sponsor | 1501 | 348
Not completed — Participant discontinued; drug related | 13 | 4
Not completed — Part. discontinued; unrelated to drug | 55 | 10
Not completed — Non-compliance with protocol | 39 | 15
Not completed — Participant moved | 40 | 12
Not completed — Participant withdrew consent | 28 | 9
Not completed — Withdrawal by Subject | 64 | 7

BASELINE CHARACTERISTICS:
Population: All Subjects as Treated Population, which consisted of all randomized participants who took at least one dose of trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | NOMAC-E2 | NETA-EE | Total
Number analyzed (Participants) | 2466 | 604 | 3070
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.2 (7.6) | 29.5 (7.7) | 29.3 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2466 | 604 | 3070
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of In-Treatment Pregnancies Per 100 Woman Years of Exposure (Pearl Index)
Description: Primary Efficacy Outcome measure for this study was contraceptive efficacy, or the prevention of in-treatment pregnancy. The total incidence of in-treatment pregnancies was expressed as the Pearl Index, which is defined as the number of in-treatment pregnancies per 100 woman-years of exposure.
Time Frame: Up to 1 year (13 cycles)
Population: Planned analysis for this primary endpoint was not performed due to early study termination.
Arm/Group | NOMAC-E2 | NETA-EE
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percentage of Participants With an Occurrence of Breakthrough Bleeding/Spotting
Description: Participants kept e-diaries to record their vaginal bleeding events. They were asked to record, on a daily basis, whether they experienced vaginal bleeding, which included BLEEDING or SPOTTING, at any time during a cycle other than normal menstruation while in the study. (This is also known as "breakthough" bleeding.) Vaginal bleeding that required >=1 pad/tampon per day was classified as BLEEDING. Vaginal bleeding that did not require a pad/tampon per day was classified as SPOTTING.
Time Frame: Up to 1 year (13 cycles)
Population: Planned analysis for this secondary endpoint was not performed due to early study termination.
Arm/Group | NOMAC-E2 | NETA-EE
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percentage of Participants With an Absence of Withdrawal Bleeding
Description: Participants kept e-diaries to record vaginal bleeding events. They were asked to record, on a daily basis, whether vaginal bleeding was present. Absence of withdrawal bleeding was defined as no bleeding/spotting during the expected bleeding period.
Time Frame: Up to 1 year (13 cycles)
Population: Planned analysis for this secondary endpoint was not performed due to early study termination.
Arm/Group | NOMAC-E2 | NETA-EE
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percentage of Participants Who Experienced At Least One Adverse Event
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study drug, whether or not it is considered related to the study drug.
Time Frame: Up to 54 weeks
Population: All Subjects as Treated Population, which consisted of all randomized participants who took at least one dose of trial medication. One treated participant in the NOMAC-E2 treatment group had incomplete data and was not included in the Safety Analyses.
Measure: Number; unit: Percentage of Participants
Arm/Group | NOMAC-E2 | NETA-EE
Number analyzed (Participants) | 2465 | 604
Percentage of Participants | 41.2 | 45.2

5. Secondary Outcome: Number of Participants Who Experience at Least One Venous or Arterial Thrombotic/Thromboembolic Event
Time Frame: Up to 54 weeks
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | NOMAC-E2 | NETA-EE
Number analyzed (Participants) | 2465 | 604
Participants | 0 | 1

6. Secondary Outcome: Change From Baseline in Body Weight
Description: Participants' body weights were measured in a consistent manner throughout the trial, using standardized equirpment. Last In-Treatment Measurement refers to a participant's end of trial visit, the timing of which differed among participants.
Time Frame: Baseline and Week 52
Population: Participants from All Subjects as Treated Population (all randomized participants who took at least one dose of trial medication) who had data available for Change from Baseline in Body Weight endpoint.
Measure: Mean (Standard Error); unit: kilograms
Arm/Group | NOMAC-E2 | NETA-EE
Number analyzed (Participants) | 2231 | 549
kilograms
  After Cycle 3 (n=2135; n=527) | 0.14 (0.14) | 0.41 (0.24)
  After Cycle 6 (n=1809; n=459) | 0.64 (0.18) | 0.29 (0.28)
  After Cycle 9 (n=1468; n=391) | 1.21 (0.23) | 0.32 (0.35)
  After Cycle 13 (n=462; n=145) | 1.57 (0.29) | 0.90 (0.46)
  Last In-Treatment Measurement (n=2231; n=549) | 1.39 (0.17) | 0.75 (0.29)

ADVERSE EVENTS:
Time Frame: Up to 54 weeks
Description: All Subjects as Treated Population, which consisted of all randomized participants who took at least one dose of trial medication. One treated participant in the NOMAC-E2 treatment group had incomplete data and was not included in the Safety Analyses.
Arm/Group | NOMAC-E2 | NETA-EE
Serious Adverse Events (participants affected / at risk) | 20/2465 | 8/604
Other Adverse Events (participants affected / at risk) | 0/2465 | 0/604
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NOMAC-E2 (N=2465) | NETA-EE (N=604)
Internal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Bacterial pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Breast cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Tubo-ovarian abscess (Infections and infestations) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic liver injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Epiphysiolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Abortion spontaneous complete (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Foetal death (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Substance abuse (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the Sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication (including slides and texts of oral or other public presentations that report any results of the trial). The Sponsor has the right to review and comment on publications, abstracts, slides, and manuscripts, as well as the data analysis and presentation.